CLINICAL TRIAL: NCT07352735
Title: Upper Extremity Sensation and Impact on Functional Use in Daily Activities in Children With Cerebral Palsy: A Comparison With Typically Developing Peer
Brief Title: Upper Extremity Sensation and Function in Children With Cerebral Palsy
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sezen Tezcan, Assist. Prof, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-ST-08
Record Dates: First submitted 2025-12-12; First posted 2026-01-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Cerebral Palsy; Sensation Disorders; Upper Extremity Dysfunction
MeSH Terms: conditions — Cerebral Palsy; Sensation Disorders | interventions — Touch

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spastic Cerebral Palsy: Individuals between the ages of 6-15 years with a diagnosis of spastic cerebral palsy
  Interventions: Diagnostic Test: Vibration Sense Assessment; Diagnostic Test: Stereognosis; Diagnostic Test: Tactile Sense; Diagnostic Test: Two Point Discrimination; Diagnostic Test: Joint position sense; Diagnostic Test: Jebsen-Taylor EHand Function Test; Other: ABILHAND-Kids survey
- Typical Developing: Typically developing individuals between the ages of 6-15
  Interventions: Diagnostic Test: Vibration Sense Assessment; Diagnostic Test: Stereognosis; Diagnostic Test: Tactile Sense; Diagnostic Test: Two Point Discrimination; Diagnostic Test: Joint position sense; Diagnostic Test: Jebsen-Taylor EHand Function Test; Other: ABILHAND-Kids survey

INTERVENTIONS:
Diagnostic Test: Vibration Sense Assessment — Vibration sense assessment with a tuning fork is based on obtaining feedback from the patient regarding the sensation of vibration by touching the vibrating tuning fork to bone or a bony prominence. The patient is asked to close their eyes, and the vibrating tuning fork is usually placed on a bone at the extremities. The tuning fork (usually 128 Hz) is struck against the hypothenar eminence of the hand or the edge of a table to vibrate. The patient is then asked to state when the vibration ceases as the tuning fork is touched to the relevant area of their body.
Diagnostic Test: Stereognosis — Participants' stereognosis sense will be assessed by placing three familiar objects (key, spoon, clothespin) and three similar matching objects (e.g., button, safety pin, pencil) in their hands. Participants will be given objects to hold and asked to identify them while blindfolded. The object will remain in the participant's hand for a maximum of 30 seconds. They will receive scores ranging from 0 to 6, first for the dominant side and then for the non-dominant side.
Diagnostic Test: Tactile Sense — The Semmes-Weinstein monofilament test is a method used to test the sense of touch in diseases that can cause various types of sensory loss. The Semmes-Weinstein Monofilament set starts with the thinnest monofilament, which should be felt at the normal level in the first stage of the test, and progresses to darker-colored monofilaments with increasing pressure. A monofilament is touched to the same area three times, and at least two of these must be correctly identified. Green indicates normal sensation, blue indicates decreased light touch sensation, purple indicates decreased protective sensation, and red indicates complete
Diagnostic Test: Two Point Discrimination — Two-point discrimination measures an individual's ability to perceive two stimulus points simultaneously. Within the scope of the study, a discriminator will be used to evaluate individuals' two-point discrimination sense. The individual will be asked to close their eyes and will be tested by moving the discriminator's index finger over their fingertip. The assessment will start at the maximum distance and will be gradually reduced until the individual can no longer distinguish between the two points. When the individual perceives the two points as one in two out of three trials, the distance will be noted in mm. To apply as equal pressure as possible, light pressure will be applied to both ends of the discriminator simultaneously.
Diagnostic Test: Joint position sense — Upper extremity proprioception will be assessed using the Joint Position Sense (JPS) test in individuals. The Angulus (DPP, USA) mobile application will be utilized as the measurement tool for this test. Participants will be positioned in a supported sitting position with the forearm in pronation and the hand placed on the table. With the participant's eyes closed, the evaluator will passively bring the wrist to an approximate $30^\circ$ extension position and hold it for 10 seconds to allow the participant to perceive the position. The wrist will then be returned to the starting (neutral) position, and the participant will be asked to actively bring their wrist to the same perceived position. This process will be repeated three times for each side. The error score will be calculated as the absolute difference between the passive target angle and the angle produced during active repositioning. The average value of the three differences will be used for the final analysis.
Diagnostic Test: Jebsen-Taylor EHand Function Test — The Jebsen-Taylor Hand Function Test (JTHFT) is a standardized and objective test of fine and gross motor hand function using tasks that mimic activities of daily living (ADL). The test consists of 7 subtests performed with the dominant and non-dominant hands. During the assessment, children will be seated in a back-supported chair with their feet flat on the floor. The writing subtest will not be administered to children who are too young to have learned to read and write. Both hands will be tested separately. Before each test item, the patient will be shown how to perform the task and will be instructed to perform the same activity first with one hand and then with the other. For each sub-item, the patient will start with the command "start" and the stopwatch will be stopped when they finish. The test completion time will be recorded for each sub-test.
Other: ABILHAND-Kids survey — The ABILHAND Kids survey will be used to assess hand dexterity, defined as the ability to manage daily activities requiring the use of the upper extremities, regardless of the strategies involved. Abilhand-Kids is a measure that can be used to assess hand skills in children with cerebral palsy. It contains 21 sub-items. The sub-items are scored as 0; cannot do, 1; has difficulty doing, and 2; does easily. The questions are usually answered by the parent, but if the child is old enough and has the appropriate cognitive level, they can also answer themselves.

SUMMARY:
This cross-sectional study was designed to evaluate upper extremity sensation in children with spastic cerebral palsy and to investigate its effect on upper extremity use in activities of daily living. Children aged 6-15 years with cerebral palsy (n=12) and typically developing peers (n=12) who volunteer to participate in the study will be included. Participants' sociodemographic data will be recorded, and upper extremity vibration sense, stereognosis, tactile sense, two-point discrimination, and joint position sense will be assessed. In the final stage, the Jebsen Taylor Hand Function Test will be administered, and parents will be asked to complete the Abilhand Kids Hand-Related Ability Scale.

DETAILED DESCRIPTION:
Recent studies have shown that sensory impairments directly affect upper extremity use. Furthermore, it has been noted that sensory functions such as stereognosis and two-point discrimination are closely related to motor skills and affect hand use in activities of daily living, that impairments in proprioceptive feedback reduce upper extremity coordination and functional task performance, and that sensory impairments limit the use of the available hand in bimanual tasks. These studies emphasize that sensory inputs form the basis for motor outputs in daily living activities and that sensory training should be prioritized in rehabilitation processes. Although the presence of sensory impairments in children with CP has been reported in the literature, the relationship between these sensory impairments and upper extremity use in activities of daily living has been addressed in a limited number of studies. In particular, the effect of senses such as vibration and stereognosis on functional outputs has not yet been sufficiently researched. This study aims to systematically examine the effect of sensory impairments on functional hand use for the first time using multidimensional sensory assessment methods. In this respect, the study will provide important and original contributions to the literature.

ELIGIBILITY:
Inclusion Criteria for Cerebral Palsy participants:

* Having a diagnosis of Cerebral Palsy
* Being between the ages of 6 and 15
* Volunteering to participate in the study

Exclusion Criteria for Cerebral Palsy participants:

* Presence of spasticity that limits active wrist movements
* Having undergone botulinum toxin or surgical procedures involving the upper extremities within the last 6 months Refusing to participate in the study

Inclusion Criteria for Typical Developing participants:

* Being between the ages of 6 and 15
* Volunteering to participate in the study

Exclusion criteria for Typical Developing participants:

* Refusing to participate in the study
* Having a history of upper extremity injury or dysfunction or mental disability

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children diagnosed with spastic cerebral palsy and typically developing peers who agreed to participate in the study and met the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Vibration Sense | through study completion, an average of 1 year
  To assess the vibration sensation of the children included in the study, a 128 Hz tuning fork (Baseline® Tuning Fork, New York, USA) will be used. In this study, participants will be seated on a table with their hips and knees at a 90-degree angle. The tuning fork will then be vibrated by tapping it against the edge of the table, and to ensure the individual feels the vibration, it will first touch their chin. The patient will then be asked to close their eyes, the tuning fork will be vibrated again by tapping it against the edge of the table, and then it will touch the dorsal part of the 1st metacarpal bone. Simultaneously, a stopwatch will be started, and the patient will be asked to state when the vibration stops, and the time will be recorded. The same procedure will be performed first on the non-dominant side and then on the dominant side. The test will be repeated 3 times, and the average of the recorded values will be taken.
stereognosis | through study completion, an average of 1 year
  In this study, individuals' stereognosia will be assessed by placing three familiar objects (key, spoon, clothespin) and three similar matching objects (e.g., button, safety pin, pencil) in their hands. Participants will be given the objects and asked to identify them with their eyes closed. The object will remain in the participant's hand for a maximum of 30 seconds. They will receive scores ranging from 0 to 6, first for the dominant side and then for the non-dominant side.
Tactile Sense | through study completion, an average of 1 year
  The Semmes-Weinstein monofilament hand kit (Fei-USA) will be used to assess individuals' tactile sensation. The test will begin with the thinnest monofilament, where the normal pressure should be felt, and progress to darker monofilaments where pressure increases. A trial test will be conducted once with eyes open and closed before the assessment to familiarize each child with the test. The monofilament will be held perpendicular to the skin and pressed against the skin until it slightly bulges. The pressure will be held for 1.5 seconds. The child will be asked if they felt the touch. Assessments will be made on the fingertips and the center of the palm.
Two-Point Discrimination | through study completion, an average of 1 year
  This study will use a discriminator (Baseline® Discrim-A-Gon 2-Point Discriminator, Fei-USA) to assess individuals' two-point discrimination sense. Individuals will be asked to close their eyes, and the discriminator will be tested by moving it over the pulp of their index finger. The assessment will begin at the maximum distance and gradually decrease until the individual can no longer distinguish between the two points. If the individual perceives the two points as one in two out of three trials, the distance will be noted in millimeters. Light pressure will be applied simultaneously to both ends of the discriminator to ensure as even pressure as possible.
Joint position sense | through study completion, an average of 1 year
  Joint position sense will be assessed using the Angulus (DPP, USA) test. With eyes closed, the participant's wrist will be passively extended to approximately 30 degrees and held for 10 seconds. Then, the wrist will be returned to the starting (neutral) position, and the participant will be asked to actively return their own wrist to the same position. This process will be repeated three times for each side. The positions achieved by the participant will be measured, and the angle difference between the passive-target position and the active-repositioning will be recorded. The difference between the target angle and the angle produced by the individual will be determined as the error score. Three measurements will be taken, and the average of the differences will be used for analysis. A 30-second rest period will be given between each trial.
Jebsen-Taylor Hand Function Test | through study completion, an average of 1 year
  The Jebsen-Taylor Hand Function Test (JTHFT) is a standardized and objective test of fine and gross motor hand function using tasks that mimic activities of daily living (ADL). The test consists of seven subtests performed with both dominant and non-dominant hands: writing, card flipping, picking up and placing small objects, stacking checkers, simulated feeding, carrying light objects, and carrying heavy objects. During the assessment, children will be seated in a chair with back support, with their feet flat on the floor. The writing subtest will not be administered as some children may not be at an age to learn to read and write. Each hand will be tested separately. Before each test item, the patient will be shown how to perform the task, instructed to perform the same activity first with one hand and then with the other. For each subtest, the patient will begin with the command "start," and the timer will stop at the end. The time taken to complete each subtest will be recorded.
Abilhand Kids | through study completion, an average of 1 year
  The Abilhand Kids questionnaire will be used to assess a child's hand dexterity, defined as their ability to manage daily activities requiring the use of the upper extremities, regardless of the strategies involved. Abilhand-Kids is a scale that can be used to assess hand dexterity in children with cerebral palsy (CP). It contains 21 sub-items. The sub-items are scored from 0; cannot, 1; has difficulty, and 2; can easily. The questions are usually answered by the parent, but the child can also answer them if they are old enough and have the appropriate cognitive level.

CONTACTS AND LOCATIONS:
Overall Officials: Sezen Tezcan, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No